CLINICAL TRIAL: NCT04221412
Title: JNJ-53718678 RSV Pre-Approval Access_Single Patient Access (SPR) for Patients Diagnosed With RSV
Brief Title: Pre-Approval Access to JNJ-53718678 for the Treatment of Respiratory Syncytial Virus (RSV) Infection in (a) Immunocompromised Adult and Pediatric Participants
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108653; 53718678RSV4001 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Syncytial Virus
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: JNJ-53718678 — JNJ-53718678 will be administered as directed by treating physician.

SUMMARY:
The purpose of this pre-approval access program is to provide treatment to immunocompromised participants with serious/life-threatening diseases or conditions (Respiratory Syncytial Virus [RSV] infection) and to collect the safety data to understand the safety profile of JNJ-53718678.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC